CLINICAL TRIAL: NCT05797454
Title: Efficacy and Accuracy of Combined Localization Versus Single Localization in Non-palpable Breast Cancer: a Prospective Randomized Control Trial.
Brief Title: Efficacy and Accuracy of Combined Localization Versus Single Localization in Non-palpable Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chang Gong, Clinical Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-129-01
Record Dates: First submitted 2023-02-26; First posted 2023-04-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Breast-conserving Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Untreated patients-combined localization (Experimental): In untreated non-palpable breast cancer patients, positioning focus use wire and marker clip at 1day before operation
  Interventions: Procedure: Wire-guided localization and marker clip localization
- Untreated patients-single localization (Active Comparator): In untreated non-palpable breast cancer patients, positioning focus use wire at 1day before operation
  Interventions: Procedure: Wire-guided localization

INTERVENTIONS:
Procedure: Wire-guided localization and marker clip localization — Positioning guide wire and marker clip in the center of the lesion
  Arms: Untreated patients-combined localization
Procedure: Wire-guided localization — Positioning guide wire in the center of the lesion
  Arms: Untreated patients-single localization

SUMMARY:
The standard method for localizing non-palpable breast cancer is currently preoperative wire-guided localization, its positive margin rate still remains around 20-50%. This study aims to compare the accuracy and efficacy of wire vs. combined breast tissue markers in localizing non-palpable breast cancer.

DETAILED DESCRIPTION:
The standard method for localizing non-palpable breast cancer is currently preoperative wire-guided localization. This study aims to compare the accuracy and efficacy of wire vs. combined breast tissue markers in localizing non-palpable breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. female patients, age≥18 year
2. A score of ≥ 2 on the Eastern Cooperative Oncology Group scale
3. Patients pathologically diagnosed with untreated breast cancer by core-needle biopsy, with histologically confirmed non-palpable in situ cancer, including pleomorphic lobular carcinoma in situ or invasive non-palpable breast cancer that required localization
4. Patients are willing to undergo breast conserving surgery and have no contraindications to breast conserving surgery.

Exclusion criteria:

1. Inflammatory breast cancer or Paget's disease
2. Breast deformities and other conditions that impact breast conservation success rate
3. Patients with contraindications to breast-conserving surgery, as well as those with systemic diseases, mental disorders, or other subjective reasons that may affect their ability to participate in the trial. Patients with severe bleeding disorders or coagulation disorders were also excluded
4. Pregnancy or lactation
5. Patients with hookwire, radioactive 125I seed or other localization techniques in the breast cancer lesions before enrollment
6. Patients with stage IV diseases or unresectable lesions in either breast
7. Patients combined with other diseases that may affect survival
8. Patients with multicentric breast cancer lesions or lesions > 5 cm in diameter on imaging examinations
9. Patients who have previously undergone radical mastectomy for ipsilateral breast cancer or chest wall radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
positive margin rate | up to 3 months
  It is defined as the proportion of patients in whom in situ or invasive carcinoma is found in the cavity margins after the first resection, including intraoperative frozen-section analysis and postoperative formalin-fixed paraffin-embedded analysis, subject to postoperative analysis.

SECONDARY OUTCOMES:
Re-operation rate | up to 3 months after first operation
  the proportion of patients which have a positive margin and requires reoperation
The proportion of breast-conserving surgery | up to 3 months after first operation
  It refers to the proportion of patients who have successfully undergone breast-conserving surgery.
IDFS | 2 years, 3 years, and 5 years
  Time from surgery to the first occurrence of local, distant disease recurrence, or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No